CLINICAL TRIAL: NCT00990717
Title: A Dose Escalation Study of NK-92 Cell Infusions in Patients With Hematological Malignancies in Relapse After Autologous Stem Cell Transplantation.
Brief Title: Safety Study Looking at the Use of a Natural Killer Cell Line Against Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP04.NK92.01
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia; Lymphoma; Myeloma; Hodgkin's Disease
Keywords: natural killer cells; leukemia; lymphoma; myeloma; Hodgkin's disease; cell therapy
MeSH Terms: conditions — Leukemia; Lymphoma; Neoplasms, Plasma Cell; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NK-92 cells (Experimental): Preparation of irradiated NK-92 cells suspended in a saline and plasma solution. NK-92 working cell bank was established from a master cell bank supplied by Conkwest Inc. (San Diego CA).
  Interventions: Biological: NK-92 cells

INTERVENTIONS:
Biological: NK-92 cells — Cells are administered as an intravenous infusion over one hour on days 1, 3 and 5 of each cycle of treatment. Patients can receive up to 6 cycles, which are administered monthly. Cell dosage is as follows:
  * Level I: 1x10^9 cells/m^2
  * Level II: 3x10^9 cells/m^2
  * Level III: 5x10^9 cells/m^2

SUMMARY:
The purpose of this study is to find out how many irradiated natural killer (NK) cells can be safely given to patients with cancer that has recurred after an autologous stem cell transplant, and to see what effects (good and bad) it has on the patient and their cancer. This research is being done because currently, there is no cure or effective treatment for blood-borne cancers when it has come back after an autologous stem cell transplant.

DETAILED DESCRIPTION:
Patients with hematological malignancies such as acute leukemia, lymphoma, Hodgkin's disease and myeloma, are generally treated initially with chemotherapy, radiotherapy or a combination of both. High dose therapy and autotransplantation are often utilized in the management of such patients, either as part of initial therapy or for treatment of relapsed disease. When a patient's cancer relapses after transplantation, the prognosis is dismal. Therapeutic options are usually limited to palliative chemotherapy and/or local radiation, and for persons with excellent performance status experimental treatments are considered on an ad hoc basis.

Much interest in the last decade has focused on the role of cellular and immunotherapy in this setting. Cancer vaccines and the administration of adoptive cellular and immunotherapy have the theoretical advantage of being non cross-reactive with previous treatments (such as radiotherapy and chemotherapy) and are currently under investigation using a variety of methodologies. NK cells comprise roughly 15% of all lymphocytes in the peripheral blood. They normally function as part of the innate immune system, which provides the body's initial response to infection and malignancy. However, patients with malignancies frequently have impaired NK cell function, as evidenced by reduced in vitro proliferative responses and reduced cytotoxic activity. The infusion of an irradiated NK cell line is appealing as it is a source of cells that can be expanded to therapeutic quantities, and retains anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Hematological malignancy (with prior histological confirmation) that has relapsed after an autologous stem cell transplant and for which there is no known curative or standard therapy. Specific hematological malignancies include acute myeloid leukemia, acute lymphoblastic leukemia, non-Hodgkin's lymphoma, Hodgkin's disease and multiple myeloma.
* Assessable disease as measured by clinical, radiological or bone marrow examinations
* ECOG performance status 0, 1 or 2
* Age ≥ 18 years
* Life expectancy greater than 12 weeks
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and University Human Experimentation Committee requirements.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: Absolute granulocytes ≥ 0.5 x 109/L, Platelets ≥ 50 x 109/L, Serum creatinine < 1.5 x upper limit of normal, Bilirubin < 1.5 x upper limit of normal, AST/ALT ≤ 3 x upper limit of normal, Calcium < 1.25 x upper limit of normal. These tests must be conducted within 7 days prior to registration.
* Must be able to come to Princess Margaret Hospital, Toronto, Canada for treatment and follow-up.

Exclusion Criteria:

* Pregnant or nursing women may not participate.
* Men or women of reproductive potential may not participate unless they agree to practice an effective method of birth control. Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to registration.
* Concurrent treatment, or treatment within 28 days of registration with other experimental drugs or anticancer therapy. Exceptions to this are: Patients who are receiving or who have received radiation therapy less than four weeks prior to study entry will not be excluded providing the volume of bone marrow treated is less than 10% and that the patient has measurable disease outside the radiation field. Hydroxyurea may be administered to patients with high white cell counts but must be discontinued at least 48 hours prior to the NK-92 cell infusions
* Patients with CNS involvement
* Known HIV, HBV or HCV infection
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular events within 3 months of registration, or psychiatric or emotional disorders.
* Patients with hypersensitivity or previous severe reactions to Allopurinol, Acetominophen or Benadryl and all available alternative medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Determine if there are any dose limiting toxicities to this therapy, as well as the maximum tolerated dose. | Day 1, 3, and 5 of each cycle

SECONDARY OUTCOMES:
Document any preliminary efficacy information from the NK-92 cell infusion. | 6 months
Assess any immune response directed against the infused NK-92 cells. | 28 days after each cycle
Determine kinetics of infused NK92 cells. | Pre-infusion, 15 min, 2h, 6h, 24h, 48h, 168h post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Armand Keating, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Klingemann HG, Martinson J. Ex vivo expansion of natural killer cells for clinical applications. Cytotherapy. 2004;6(1):15-22. doi: 10.1080/14653240310004548. PMID 14985163
- [Background] Gong JH, Maki G, Klingemann HG. Characterization of a human cell line (NK-92) with phenotypical and functional characteristics of activated natural killer cells. Leukemia. 1994 Apr;8(4):652-8. PMID 8152260
- [Background] Tam YK, Miyagawa B, Ho VC, Klingemann HG. Immunotherapy of malignant melanoma in a SCID mouse model using the highly cytotoxic natural killer cell line NK-92. J Hematother. 1999 Jun;8(3):281-90. doi: 10.1089/106161299320316. PMID 10417052
- [Background] Maki G, Tam YK, Berkahn L, Klingemann HG. Ex vivo purging with NK-92 prior to autografting for chronic myelogenous leukemia. Bone Marrow Transplant. 2003 Jun;31(12):1119-25. doi: 10.1038/sj.bmt.1704117. PMID 12796791